CLINICAL TRIAL: NCT05677152
Title: Influence of Zoledronic Acid on Healing After Arthroscopic Repair of Chronic Rotator Cuff Lesions - A Prospective, Randomized, Placebo-controlled Phase II Trial
Brief Title: Influence of an Anti-osteoporotic Drug on Healing After Surgical Repair of Chronic Rotator Cuff Lesions of the Shoulder
Acronym: ZORRO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AUVA Traumazentrum Vienna Site UKH Meidling (Other)
Collaborators: Ludwig Boltzmann Institute for Traumatology - The research center in cooperation with AUVA (Other Government)
Responsible Party: Principal Investigator, Jakob Schanda, Principal Investigator, AUVA Trauma Center Meidling
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZORRO
Record Dates: First submitted 2022-06-02; First posted 2023-01-10 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Orthopedics; Traumatology
Keywords: zoledronic acid; chronic rotator cuff tears; arthroscopic repair

STUDY DESIGN:
Intervention Model Description: placebo controlled trial (Zoledronic acid versus Placebo), randomized,
  2 Teams: unblinded and blinded
Who Masked: Participant, Investigator
Masking Description: In this trial, zoledronic acid or placebo will be administered once immediately before arthroscopic rotator cuff repair.
  Randomization will take place. immediately before surgery by the anesthesiologist using sealed envelopes. To simplify the study procedure, zoledronic acid 5 mg (Aclasta®), administered as single intravenous infusion (verum) or sodium chloride (physiological saline solution 0.9%), administered as single intravenous infusion (placebo) will be administered preoperatively by the anesthesiologist after induction of anesthesia. Thereby, patients and surgeons are blinded to the randomization process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zoledronic Acid (Active Comparator): zoledronic acid 5 mg (Aclasta®) administered as single intravenous infusion (100 ml): Verum
  Interventions: Drug: Intravenous Infusion of Aclasta®
- physiological saline solution 0.9% (Placebo Comparator): Sodium chloride (physiological saline solution 0.9%) administered as single intravenous infusion (100 ml): Placebo
  Interventions: Drug: Intravenous Infusion of Aclasta®

INTERVENTIONS:
Drug: Intravenous Infusion of Aclasta® — Intravenous Infusion of Aclasta® (Verum) or physiological saline solution 0.9% (Placebo)

SUMMARY:
This is a prospective, single-center, placebo-controlled, non-comparative, phase II study to evaluate the influence of an adjuvant, intravenous therapy with zoledronic acid (single dose) on healing after arthroscopic repair of chronic rotator cuff tears.

The study including its financial support was approved by the medical director of the General Accident Insurance Institution (AUVA) , Dr. Roland Frank.

Hypothesis to prove: Adjuvant intravenous therapy with zoledronic acid does improve tendon healing after arthroscopic reconstruction of chronic rotator cuff tears compared to a control group without adjuvant therapy with zoledronic acid.,

ELIGIBILITY:
Inclusion Criteria

* Age between 50 and 70 years
* Magnetic resonance imaging verified rotator cuff tear (within 6 month prior to surgery)
* Rupture size with a maximum diameter of 3 cm
* Willingness to participate in the study
* Willingness to participate in a unified physiotherapy with use of a shoulder abduction pad for four weeks postoperativel

Exclusion Criteria:

* Patients younger than 50 or older than 70 years of age
* Pregnancy
* Known allergy to zoledronic acid or other components of the medicinal product
* Previous fracture of the affected shoulder
* Previous surgery of the affected shoulder
* Previous or existing bacterial infection of the affected shoulder
* Rupture of more than two tendons in the affected shoulder (massive rotator cuff tear)
* Isolated subscapularis tendon tear
* Presence of glenohumeral osteoarthritis (Hamada type 3 or higher)
* Diabetes mellitus (fasting glucose ≥ 126 mg/dl, HbA1C ≥ ZORRO Version Draft1.0/09.05.2022 Page 6 of 42 6.5%)
* Malignant tumor disease
* Pathological dental status
* Known disease that interferes with bone metabolism
* Concomitant diseases that do not permit general anesthesia
* Previous therapy with anti-osteoporotic drugs (bisphosphonates, denosumab, teriparatide)
* Epilepsy
* Claustrophobia
* Chronic alcohol abuse
* Drug abuse

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Tendon integrity of the rotator cuff by means of magnetic resonance imaging. | 8 years
  postoperative anatomically regular tendon thickness comparable to an intact tendon.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Schanda, DDr., Principal Investigator — AUVA Traumazentrum Vienna Site UKH Meidling
Locations (1):
- Jakob Schanda, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schanda JE, Ullrich R, Boesmueller S, Mittermayr R, Bruell T, Hexel M, Heuberer PR, Woisetschlaeger G, Neuper OM, Redl H, Grillari J, Fialka C. Intraoperative Zoledronic Acid for Arthroscopic Rotator Cuff Repair: Short-Term Results From a Prospective, Randomized, Placebo-Controlled Phase II Trial. Am J Sports Med. 2026 Jan 18:3635465251399167. doi: 10.1177/03635465251399167. Online ahead of print. PMID 41549490